CLINICAL TRIAL: NCT03655145
Title: Randomized Prospective Phase III Clinical Trial Comparing HLA 10/10 Matched Unrelated Donor and Haploidentical Allogenic Hematopoietic Stem Cell Transplantation After Myeloablative Conditioning Regimen
Brief Title: HLA 10/10 Matched Unrelated Donor vs Haploidentical Allogenic Hematopoietic Stem Cell Transplantation
Acronym: MacHaploMud
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AOM 17030
Record Dates: First submitted 2018-06-06; First posted 2018-08-31 (Actual); Last update posted 2018-08-31 (Actual); Status verified 2018-05

CONDITIONS: Acute Myeloid Leukemia; Acute Lymphoblastic Leukemia; Myeloproliferative Syndromes; Myelodysplastic Syndromes
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Myelodysplastic Syndromes

STUDY DESIGN:
Intervention Model Description: Randomized prospective Phase III clinical trial comparing HLA 10/10 matched unrelated donor (standard arm) and haploidentical allogeneic hematopoietic stem cell transplantation (experimental arm) after myeloablative conditioning regimen
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Haploidentical donor stem cell transplantation (Experimental): The stem cell source will be bone marrow for haploidentical transplantation.The bone marrow collection is carried out according to the practice of each centre with a minimal target dose of 3x108 TNC/kg.
  Interventions: Other: Haplo donor stem cell transplantation
- HLA 10/10 MUD stem cell transplantation (Active Comparator): The stem cell source will be peripheral blood stem cell for HLA-matched unrelated transplantation.Peripheral blood stem cell (PBSC) for HLA-matched unrelated SCT will be mobilized by G-CSF (Neupogen®) administered to the donor from Day-4 to Day-1 subcutaneously (10µg/kg/day) with the minimal target dose of 4.106 CD34+ cells/kg.
  Interventions: Other: HLA 10/10 MUD stem cell transplantation

INTERVENTIONS:
Other: Haplo donor stem cell transplantation — The algorithm for selection of haploidentical donor has been defined by the french society for stem cell transplantation The stem cell source will be bone marrow for haploidentical transplantation.The bone marrow collection is carried out according to the practice of each centre with a minimal target dose of 3x108 TNC/kg.
  Arms: Haploidentical donor stem cell transplantation
Other: HLA 10/10 MUD stem cell transplantation — HLA 10/10 matched unrelated donor myeloablative transplantation
  Arms: HLA 10/10 MUD stem cell transplantation

SUMMARY:
The MAC-HAPLO-MUD trial is a randomized prospective phase III trial comparing HLA 10/10 matched unrelated donor and haploidentical allogeneic hematopoietic stem cell transplantation after myeloablative conditioning regimen in patients, age 15 years or older, with Acute Myeloid Leukemia (AML) or Acute Lymphoblastic Leukemia (ALL) or Myeloproliferative Syndrome (SMP) or Myelodysplastic Syndromes (SMD) and requiring allogeneic hematopoietic stem cell transplantation. Primary endpoint is the 1-year progression free survival without acute grade II-IV GvHD and without moderate and severe chronic GvHD.

DETAILED DESCRIPTION:
An unrelated adult donor who is HLA-matched to the recipient at the allele-level (at HLA-A, -B, -C, -DQB1 and -DRB1) is considered the best choice in the absence of an HLA-matched sibling for patients needing hematopoietic stem cell transplantation (SCT).

However, using matched unrelated donors (MUD) is limited by (1) a prolonged time to identify and schedule donation for some MUD allowing some patients to relapse before transplantation can be performed, and (2) limited availability of fully HLA-MUD for the non-Caucasian population.

Alternative donors are used for transplantation in patients without a fully-MUD including single HLA mismatched unrelated donor, unrelated umbilical cord blood and grafts from haploidentical related donors but are associated with higher non-relapse mortality and delayed immune reconstitution.

A more recent strategy for haploidentical (haplo) related donor SCT (haplo-SCT) has improved dramatically outcomes using T-cell replete grafts with administration of post-transplantation cyclophosphamide (PTCy).

From retrospective studies, haplo-SCT with PTCy are associated with similar overall and progression-free survivals as with MUD stem cell transplantation (MUD-SCT), but with lower rates of toxicity and graft versus host disease (GvHD), and thus potentially better results than MUD-SCT after reduced intensity conditioning (RIC) regimen. Haplo-SCT with PTCy is thus highly discussed nowadays motivating prospective trials to confirm the benefit of this procedure.

In the setting of a myeloablative conditioning (MAC) regimen in adults with high risk hematological malignancies, few retrospective non-controlled registry studies recently suggest that outcomes after haplo-SCT using PTCy approach might also be superior in terms of GVHD free survival to that after MUD stem cell transplantation (MUD-SCT).

The investigators propose to address this question, in a randomized prospective phase III clinical trial comparing HLA 10/10 MUD and haplo-SCT after MAC regimen. The stem cell source will be bone marrow for haploidentical SCT and peripheral blood stem cell (PBSC) for HLA-matched unrelated transplantation.

The primary endpoint is the 1-year progression free survival without acute grade II-IV GvHD and without moderate and severe chronic GvHD.

ELIGIBILITY:
Inclusion Criteria:

* With AML/ALL/SMD/SMP requiring allogeneic stem cell transplantation
* In complete response (CR) for AML/ALL or in CR, or partial response (PR) or non pre-treated for SMD/SMP *
* Without a HLA matched related donor available
* With a good probability to have a HLA-10/10 matched donor available (the patient needs to have at least 5 MUD identified within the book "BMDW (Bone Marrow Donors Worldwide)"
* With identification of a haploidentical donor (brother, sister, parents, adult children or cousin)
* Absence of donor specific antibody (DSA) detected in the patient with a MFI ≥ 2000 (antibodies directed towards the distinct haplotype between donor and recipient)

With usual criteria for hematopoietic stem cell transplant (HSCT):

* Eastern Cooperative Oncology Group (ECOG) ≤ 2
* No severe and uncontrolled infection
* Cardiac function compatible with high dose of cyclophosphamide
* Adequate organ function: aspartate transaminase (ASAT) and alanine aminotransferase (ALAT) ≤ 2N, total bilirubin ≤ 1.5N, creatinine clearance ≥30ml/min (except if those abnormalities are linked to the hematological disease)

  * With health insurance coverage
  * Understand informed consent or optimal treatment and follow-up
  * Contraception methods must be prescribed during all the duration of the research and using effective contraceptive methods during treatment and within 12 months for women and 6 months for men after the last dose of cyclophosphamide
  * Having signed a written informed consent (2 parents for patients aged less than 18)

Exclusion Criteria:

* Presence of donor specific antibody (DSA) with a MFI ≥ 2000 detected in the patient
* History of Cancer in the last 5 years (except basal cell carcinoma of the skin or "in situ" carcinoma of the cervix)
* Uncontrolled infection
* Seropositivity for HIV or HTLV-1 or active hepatitis B or C defined by a positive polymerase chain reaction (PCR) hepatitis B virus (HBV) or hepatitis C virus (HCV) and hepatic cytolysis due to HBV
* Yellow fever vaccine within 2 months before transplantation
* Uncontrolled coronary insufficiency, recent myocardial infarction <6 month, current manifestations of heart failure, uncontrolled cardiac rhythm disorders, ventricular ejection fraction <50%
* Heart failure according to New York Heart Association (NYHA) (II or more)
* Urinary tract obstruction
* Contraindications to treatments used during the research
* Preexisting acute hemorrhagic cystitis
* Renal failure with creatinine clearance <30ml / min
* Pregnancy ( β- human chorionic gonadotropin (β-HCG positive)) or breast-feeding
* Any debilitating medical or psychiatric illness which would preclude the realization of the SCT or the understanding of the protocol
* Under protection by law (tutorship or curatorship)
* Unwilling or unable to comply with the protocol

Ages: 15 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 344 (Estimated)
Dates: Start 2018-08 (Estimated); Primary Completion 2019-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Progression free survival, without acute grade II-IV GvHD and without moderate and severe chronic GvHD. | 12 months
  One year progression free survival, without acute grade II-IV GvHD and without moderate and severe chronic GvHD.
  -Relapse evaluation:
  For myeloid malignancies, the relapse will be defined by the reappearance of leukemic cells after SCT.
  For ALL, the relapse will be defined by: the reappearance of leukemic cells after SCT and/or an increase of at least 50 % of the smallest measure of any lymphnode considered abnormal in the pre-transplantation period for patients in partial response and in non-responders and/or the appearance of any new lesion in comparison with the pre-transplantation period evaluation.
  - GvHD evaluation:
  Grading of acute GVHD will be performed according to the classification of Glusckberg.
  Grading of chronic GVHD will be performed according to the NIH classification.

SECONDARY OUTCOMES:
Time interval between indication of stem cell transplantation (SCT) and transplant | 24 months
Engraftment | at 24 months
  Engraftment: at least 3 consecutive days with neutrophils > 0.5 G/L, with platelets > 20 G/L
Numbers of neutrophils | at 1 month
  Absolute numbers of neutrophils
Numbers of platelets | at 1 month
  Absolute numbers of platelets
Numbers of neutrophils | at 2 months
  Absolute numbers of neutrophils
Numbers of platelets | at 2 months
  Absolute numbers of platelets
Numbers of neutrophils | at 3 months
  Absolute numbers of neutrophils
Numbers of platelets | at 3 months
  Absolute numbers of platelets
Numbers of neutrophils | at 6 months
  Absolute numbers of neutrophils
Numbers of platelets | at 6 months
  Absolute numbers of platelets
Numbers of neutrophils | at 12 months
  Absolute numbers of neutrophils
Numbers of platelets | at 12 months
  Absolute numbers of platelets
Numbers of neutrophils | at 24 months
  Absolute numbers of neutrophils
Numbers of platelets | at 24 months
  Absolute numbers of platelets
Use of growth factors | at 12 months
  Use of growth factors for poor hematopoietic reconstitution
Immune reconstitution | at 1 month post transplantation
  Immune reconstitution by analyzing T, B, Natural Killer (NK), regulatory T cell levels in the peripheral blood
Immune reconstitution | at 3 months post transplantation
  Immune reconstitution by analyzing T, B, NK, regulatory T cell levels in the peripheral blood
Immune reconstitution | at 6 months post transplantation
  Immune reconstitution by analyzing T, B, NK, regulatory T cell levels in the peripheral blood
Immune reconstitution | at 12 months post transplantation
  Immune reconstitution by analyzing T, B, NK, regulatory T cell levels in the peripheral blood
Immune reconstitution | at 24 months post transplantation
  Immune reconstitution by analyzing T, B, NK, regulatory T cell levels in the peripheral blood
Iron overload estimation | at 1 month
Iron overload estimation | at 3 months
Iron overload estimation | at 6 months
Iron overload estimation | at 12 months
Iron overload estimation | at 24 months
Chimerism | at 1 month
Chimerism | at 3 months
Chimerism | at 6 months
Chimerism | at 12 months
Acute GvHD | at 24 months
  Incidence of acute GvHD
First line treatment | 24 months
Response to steroids | 24 months
Treatment courses for refractory aGVHD | 24 months
Relapse | 24 months
  Incidence of relapse
Progression free survival | 24 months
Severe infections (CTAE grade 3-4) | 12 months
Cytomegalovirus (CMV) | 12 months
  Incidence of CMV
Epstein-Barr virus (EBV) | 12 months
  Incidence of EBV reactivation
Veno-occlusive disease (VOD) | 3 months
  Incidence of veno-occlusive disease
Severity of veno-occlusive disease (VOD) | 3 months
  Severity of veno-occlusive disease. VOD severity will be assessed using new EBMT criteria (Mohty et al., 2016). EBMT criteria for grading VOD severity in adult patients are based on the level of bilirubin and its rate of change, liver function (transaminase), weight increase, renal function and the kinetic of their onset (Mohty et al., 2016). This grading system is divided into five categories as following: mild, moderate; severe, very severe; and death.
  Mohty M., Malard F., Abecassis M., Aerts E., Alaskar AS. et al. (2016). Revised diagnosis and severity criteria for sinusoidal obstruction syndrome/veno-occlusive disease in adult patients: a new classification from the European Society for Blood and Marrow Transplantation. Bone Marrow Transplantation 51,906-912.
Cardiac toxicities | 12 months
  Incidence of cardiac toxicities
Non-relapse mortality | 12 months
Overall survival | 24 months
  Time between death and inclusion
Quality of life post transplantation: EORTC QLQ-C30- v3 | 1 week post-transplantation
  Quality of life evaluated using questionnaire "European Organization for Research and Treatment of Cancer Quality of Life Questionnaire" (EORTC QLQ-C30- v3). The QLQ-C30 is composed of both multi-item scales and single-item measures. These include five functional scales, three symptom scales, a global health status / QoL scale, and six single items. Each of the multi-item scales includes a different set of items - no item occurs in more than one scale. All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level. A high score for a functional scale represents a high/healthy level of functioning. A high score for the global health status/ QoL represents a high QoL and a high score for a symptom scale/item represents a high level of symptomatology/problems.
  EORTC QLQ-C30 Scoring Manual. Fayers PM et al. on behalf of the EORTC Quality of Life Group. EORTC, 2001. ISBN: 2-9300.
Quality of life at 3 months: EORTC QLQ-C30- v3 | 3 months
  Quality of life evaluated using questionnaire "European Organization for Research and Treatment of Cancer Quality of Life Questionnaire" (EORTC QLQ-C30- v3). The QLQ-C30 is composed of both multi-item scales and single-item measures. These include five functional scales, three symptom scales, a global health status / QoL scale, and six single items. Each of the multi-item scales includes a different set of items - no item occurs in more than one scale. All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level. A high score for a functional scale represents a high/healthy level of functioning. A high score for the global health status/ QoL represents a high QoL and a high score for a symptom scale/item represents a high level of symptomatology/problems.
  EORTC QLQ-C30 Scoring Manual. Fayers PM et al. on behalf of the EORTC Quality of Life Group. EORTC, 2001. ISBN: 2-9300.
Quality of life at 6 months: EORTC QLQ-C30- v3 | 6 months
  Quality of life evaluated using questionnaire "European Organization for Research and Treatment of Cancer Quality of Life Questionnaire" (EORTC QLQ-C30- v3). The QLQ-C30 is composed of both multi-item scales and single-item measures. These include five functional scales, three symptom scales, a global health status / QoL scale, and six single items. Each of the multi-item scales includes a different set of items - no item occurs in more than one scale. All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level. A high score for a functional scale represents a high/healthy level of functioning. A high score for the global health status/ QoL represents a high QoL and a high score for a symptom scale/item represents a high level of symptomatology/problems.
  EORTC QLQ-C30 Scoring Manual. Fayers PM et al. on behalf of the EORTC Quality of Life Group. EORTC, 2001. ISBN: 2-9300.
Quality of life at 12 months: EORTC QLQ-C30- v3 | 12 months
  Quality of life evaluated using questionnaire "European Organization for Research and Treatment of Cancer Quality of Life Questionnaire" (EORTC QLQ-C30- v3). The QLQ-C30 is composed of both multi-item scales and single-item measures. These include five functional scales, three symptom scales, a global health status / QoL scale, and six single items. Each of the multi-item scales includes a different set of items - no item occurs in more than one scale. All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level. A high score for a functional scale represents a high/healthy level of functioning. A high score for the global health status/ QoL represents a high QoL and a high score for a symptom scale/item represents a high level of symptomatology/problems.
  EORTC QLQ-C30 Scoring Manual. Fayers PM et al. on behalf of the EORTC Quality of Life Group. EORTC, 2001. ISBN: 2-9300.
Quality of life at 24 months: EORTC QLQ-C30- v3 | 24 months
  Quality of life evaluated using questionnaire "European Organization for Research and Treatment of Cancer Quality of Life Questionnaire" (EORTC QLQ-C30- v3). The QLQ-C30 is composed of both multi-item scales and single-item measures. These include five functional scales, three symptom scales, a global health status / QoL scale, and six single items. Each of the multi-item scales includes a different set of items - no item occurs in more than one scale. All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level. A high score for a functional scale represents a high/healthy level of functioning. A high score for the global health status/ QoL represents a high QoL and a high score for a symptom scale/item represents a high level of symptomatology/problems.
  EORTC QLQ-C30 Scoring Manual. Fayers PM et al. on behalf of the EORTC Quality of Life Group. EORTC, 2001. ISBN: 2-9300.
Number of new days of hospitalization after the hospitalization for transplantation | at 24 months

IPD SHARING:
Plan to Share IPD: Undecided